CLINICAL TRIAL: NCT01747083
Title: A Randomized, Open Label, Single Dose, Crossover Study to Investigate Food-effect Bioavailability of FDC(Gemigliptin/Metformin HCl Sustained Release) 50/1000mg(25/500mg x 2tablets)Under Fed and Fasting Conditions in Healthy Male Volunteers
Brief Title: Food-Effect Bioavailability Study of FDC(Gemigliptin/Metformin HCl Sustained Release) 50/1000mg(25/500mg x 2tablets)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LG-DMCL003
Record Dates: First submitted 2012-11-30; First posted 2012-12-11 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- A (Experimental): FDC(gemigliptin/metformin HCl sustained release 50/1000mg(25/500mgx2tablets))under fasting condition
  Interventions: Drug: FDC(gemigliptin/metformin HCl sustained release 50/1000mg(25/500mg x 2tablets))
- B (Experimental): FDC(gemigliptin/metformin HCl sustained release 50/1000mg(25/500mgx2tablets))under fed condition
  Interventions: Drug: FDC(gemigliptin/metformin HCl sustained release 50/1000mg(25/500mg x 2tablets))

INTERVENTIONS:
Drug: FDC(gemigliptin/metformin HCl sustained release 50/1000mg(25/500mg x 2tablets))

SUMMARY:
This study is designed to investigate the food-effects on FDC(gemigliptin/metformin HCl sustained release) 50/1000mg(25/500mg x 2tablets)

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45, healthy male subjects(at screening)
* BMI between 19.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(Aspirin, antibiotics)
* Subject who already participated in other trials in 90 days
* Subject who had whole blood donation in 60 days, or component blood donation in 30 days or transfusion in 30 days currently.
* Smokers.(but, if the subject did'nt smoke in 3months, can participate the trial)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
AUClast | up to 48 h post-dose
  To evaluate AUClast of gemigliptin and metformin
Cmax | up to 48 h post-dose
  TO evaluate Cmax of gemigliptin and metformin

SECONDARY OUTCOMES:
AUCinf | up to 48 h post-dose
  To evaluate AUCinf of gemigliptin,metformin and LC15-0636(active metabolite of gemigliptin)
Tmax | up to 48h post-dose
  To evaluate Tmax of gemigliptin, metformin and LC15-0636(active metabolite of gemigliptim)
t1/2 | up to 48 h post-dose
  To evaluate t1/2 of gemigliptin, metformin and LC15-0636(active metabolite of gemigliptim)
Cmax | up to 48h post-dose
  To evaluate Cmax of LC15-0636(active metabolite of gemigliptim)
AUClast | up to 48h post-dose
  To evaluate AUClast of LC15-0636(active metabolite of gemigliptim)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea